CLINICAL TRIAL: NCT05397821
Title: The Optimal Method for Ureter Implantation in Pediatric Kidney Transplantation
Brief Title: Pediatric Kidney Transplantation, Ureteroneocystostomy Techniques
Acronym: TUIKIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 112452
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Kidney Transplant; Complications; Kidney Transplant Infection; Kidney Transplant Failure and Rejection
Keywords: Kidney transplantation; Pediatrics
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radboudumc recipients: NTX performed with a refluxing technique
  Interventions: Procedure: UNC technique
- Winsconsin recipients: NTX performed with a non-refluxing technique
  Interventions: Procedure: UNC technique

INTERVENTIONS:
Procedure: UNC technique — In general, UNC techniques can be divided in being either intravesical or extravesical and refluxing or non-refluxing

SUMMARY:
In this study the researchers want to retrospectively compare non-refluxing ureteroneocystostomy (UNC techniques to reflux UNC techniques in paediatric kidney recipients with regard to urinary tract infections and uteral obstruction.

DETAILED DESCRIPTION:
Multi-center retrospective study and survey on clinical practice among different urologists. The researchers will retrospectively study data on patients that received their kidney graft between 1994-2018 in either Radboudumc or UW Health University Hospital in Winsconsin.

Additionally, all urologist currently employed at those hospitals will be asked to fill in a survey on preferences in UNC techniques and suture material.

ELIGIBILITY:
Inclusion Criteria:

* received kidney graft in the participating centres at an age <19
* received kidney graft between 1994-2018
* follow-up data of at least 1 year

Exclusion Criteria:

- Loss of follow up < 1 year

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric kidney recipients that were transplanted between 1994-2018 in either Radboudumc or Winconsin University
Sampling Method: Non-Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infections | 25 year
  Number of urinary tract infections (with fever)
Ureteral obstruction | 25 year
  Number of ureteral obstruction needing intervention

SECONDARY OUTCOMES:
Graft survival | 25 years
  Percentage of patients with a functioning graft

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Lamers, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, CSR
Time Frame: 25 year
Access Criteria: well written request